CLINICAL TRIAL: NCT00003057
Title: Randomized Trial of High-Dose Versus Conventional Dose Octreotide Acetate Versus Loperamide in the Treatment of Chemotherpay-Related Diarrhea in Patients With Colorectal Cancer
Brief Title: Octreotide Compared With Loperamide Hydrochloride for Chemotherapy-Related Diarrhea in Patients With Colorectal Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); SWOG Cancer Research Network (Network); Cancer and Leukemia Group B (Network)
Allocation: Randomized | Purpose: Supportive Care
Other Study IDs: CDR0000065713; E-E1295; CLB-9770; SWOG-E1295; NCI-P97-0081
Record Dates: First submitted 1999-11-01; First posted 2004-07-19 (Estimated); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Colorectal Cancer; Diarrhea
Keywords: colon cancer; rectal cancer; diarrhea
MeSH Terms: conditions — Colorectal Neoplasms; Diarrhea; Colonic Neoplasms; Rectal Neoplasms | interventions — Loperamide; Octreotide

INTERVENTIONS:
Drug: loperamide hydrochloride
Drug: octreotide acetate

SUMMARY:
RATIONALE: Drugs such as octreotide and loperamide hydrochloride use different ways to relieve the diarrhea caused by chemotherapy.

PURPOSE: Randomized phase III trial to compare the effectiveness of octreotide with loperamide hydrochloride for the treatment of chemotherapy-related diarrhea in patients who have colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the safety and efficacy of octreotide acetate versus conventional therapy with loperamide hydrochloride for chemotherapy related diarrhea in patients with advanced colorectal malignancies undergoing chemotherapy with fluorouracil or fluorouracil based regimens.

OUTLINE: This is a prospective, randomized, parallel, open label, multicenter study. Patients are stratified by therapy, grade of diarrhea, and prior use of loperamide hydrochloride or octreotide acetate. Patients undergo 1 of 3 treatments. Patients receive either low doses of octreotide (arm A) or high doses of octreotide (arm B) subcutaneously 3 times daily for 5 days. Patients in arm C receive oral doses of loperamide following each unformed stool for 5 days. A diary is completed by patients to record medications and bowel history. Treatment continues if diarrhea persists beyond day 5, but will be considered a treatment failure. If diarrhea continues to worsen, patients are removed from study. All patients are followed for 24 days.

PROJECTED ACCRUAL: This study will accrue a total of 500 patients.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed colorectal carcinoma At least grade 2 diarrhea as a consequence of chemotherapy

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Not specified Renal: Not specified Other: Concurrent enrollment into SWOG-9420 protocol allowed No sensitivity to octreotide acetate or loperamide hydrochloride Eligible if less than 24 hours since prior loperamide or octreotide and no resolution of diarrhea Not pregnant or lactating Effective contraception required of fertile patients Not HIV positive No idiopathic ulcerative colitis or Crohn's disease, acute stool culture positive bacterial colitis, pseudomembranous colitis, short bowel syndrome, enteroenteric fistulae, chronic pancreatitis, ischemic bowel disease, or gastrointestinal disorders known to cause diarrhea Absence of definitive culture results required

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: Prior chemotherapy with a fluoropyrimidine alone or in combination with an accepted modulating agent (leucovorin, levamisole, methotrexate, interferon, PALA, or hydroxyurea) required Prior chemotherapy with uracil mustard and tegafur (UFT) allowed No concurrent chemotherapy allowed during study Endocrine therapy: Not specified Radiotherapy: No whole pelvic or abdominal radiation therapy allowed Surgery: No colectomy, coloanal anastamosis, abdominoperineal resection, or colostomy allowed Other: No antidiarrheal agents (e.g., diphenoxylate hydrochloride, elixir paregoric, opium tincture or tincture of belladonna, or kaolin) during study No cyclosporine allowed

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 1997-03-26 (Actual); Primary Completion 2000-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Wadler, MD, Study Chair — Albert Einstein College of Medicine; Mace L. Rothenberg, MD, FACP, Study Chair — Vanderbilt-Ingram Cancer Center; Bhoomi Mehrotra, MD, Study Chair — Long Island Jewish Medical Center
Locations (33):
- United States (33):
  - University of California San Diego Cancer Center, La Jolla, California
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - CCOP - Christiana Care Health Services, Wilmington, Delaware
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - University of Illinois at Chicago Health Sciences Center, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Marlene & Stewart Greenebaum Cancer Center, University of Maryland, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - Ellis Fischel Cancer Center - Columbia, Columbia, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Norris Cotton Cancer Center, Lebanon, New Hampshire
  - CCOP - North Shore University Hospital, Manhasset, New York
  - North Shore University Hospital, Manhasset, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - New York Presbyterian Hospital - Cornell Campus, New York, New York
  - Mount Sinai Medical Center, NY, New York, New York
  - CCOP - Syracuse Hematology-Oncology Associates of Central New York, P.C., Syracuse, New York
  - State University of New York - Upstate Medical University, Syracuse, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - CCOP - Southeast Cancer Control Consortium, Winston-Salem, North Carolina
  - Comprehensive Cancer Center of Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Tennessee, Memphis Cancer Center, Memphis, Tennessee
  - Vermont Cancer Center, Burlington, Vermont
  - MBCCOP - Massey Cancer Center, Richmond, Virginia